CLINICAL TRIAL: NCT02606812
Title: Effect of Food Consumption on microRNA Related to Metabolic Syndrome. A Randomized Clinical Trial
Brief Title: Effect of Food Consumption on microRNA Related to Metabolic Syndrome
Acronym: EFCMRNAMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Juárez Autónoma de Tabasco (Other)
Responsible Party: Principal Investigator, JUAN MANUEL MUÑOZ CANO, M. en C., Universidad Juárez Autónoma de Tabasco
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UniversidadJAT
Record Dates: First submitted 2015-10-28; First posted 2015-11-17 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional-food (Experimental): During the 3 months, a dish containing traditional food will be provided 5 days per week. The food will contain an average of 600 Kcal, ≤ 50 mg of cholesterol, ≥ 10 g of fiber, ≥ 130 g of vegetables, and ≤ de 200 mg of sodium. Each dish will be accompanied with 3 standard-sized corn tortillas.
  Interventions: Dietary Supplement: Traditional-food
- Control (No Intervention): Is the group who will intake the cafeteria fast food. The control group will receive habitually consumed fast food provided by the cafeteria of the campus at a similar caloric proportion.

INTERVENTIONS:
Dietary Supplement: Traditional-food — Intake of ethnic local food
  Arms: Traditional-food

SUMMARY:
The objective of the Project is to assess the effect of traditional food on the expression of micro-ribonucleic acid (miRNA), which regulate genes related to glucose metabolism. It will be a randomized experimental research. The research hypothesis is that consumption of traditional food will resolve biomarkers of glucose-related anomalies. Students of The Academic Division of Health Sciences (DACS for its initials in Spanish) will be invited to participate and they will be divided randomly in two groups. The experimental group will receive daily, five days per week, during three months, a lunch based on traditional Mesoamerican food emphasizing local produce. The experimental group will be provided an equivalent ratio of fast food from the school cafeterias. In both groups, at the start and end of the protocol, values of lipid, glucose, reactive protein C, alanine aminotransferase, and glycosylated hemoglobin profiles will be determined through spectrophotometric methods. The levels of expression of five miARN involved in regulating genes related to glucose metabolism (miR-320, miR-33a/b, miR-145, miR-335, and miR-124a) will be determined also by means of PCR amplification techniques. Statistical analyses will be based on two-way ANOVA, with a Dunnet's test procedure to find significance in measurements; significance will be set at p ≤ 0.05.

DETAILED DESCRIPTION:
Study design. This is a randomized study. Freshman students at Universidad Juárez Autónoma de Tabasco (UJAT) are subjected to clinical laboratory tests as part of their enrollment process to the University. Fifty women will be invited to participate, because DACS' enrollment is predominated by women. Blood samples will be taken for clinical and molecular analyses at the start and end of the protocol (three months). Anthropometric measurements will be taken also at the start and end of the study. During the 3 months, a dish containing traditional food will be provided 5 days per week. The food will contain an average of 600 Kcal, ≤ 50 mg of cholesterol, ≥ 10 g of fiber, ≥ 130 g of vegetables, and ≤ de 200 mg of sodium. Each dish will be accompanied with 3 standard-sized corn tortillas. The control group will receive habitually consumed fast food provided by the cafeteria of the campus at a similar caloric proportion (Muñoz et al., in press)

Anthropometrics. To determine the body mass index (BMI), according to World Health Organization (2011) guidelines, a clinical balance with a stadiometer (Básculas Nuevo León®, Mexico) with a weighing capacity of 200 kg will be used. The balance will be calibrated daily during the whole time of students' recruitment. The BMI will be calculated according to the Mexican standard NOM-043-SSA2-2011 (2012). To measure hip and waist perimeters, millimetric non-extensible fiber glass tapes will be used, with a length of 1.80 m and a width of 1 cm (Vitamex® Mexico). For the population of this region, the desirable hip measure for women is of 80 cm and of 90 cm for men (WHO, 2011). The waist/hip ratio (WHR) is calculated by dividing the waist perimeter by the hip perimeter, where a value of 0.85 for women and of 0.90 for men are considered the cut-off limits (He et al., 2009). The waist-to-height ratio (WHtR) is calculated by dividing the waist measurement by that of height, where a value below 0.5 is considered desirable (WHO, 2011).

Biochemical parameters. Blood samples from participants will be procured by personnel of the clinical analyses laboratory of UJAT after a 12-hour fasting period. Sterile equipment will be used and blood will be collected in Vacutainer® Serum tubes (BectonDickinson, Franklin Lakes, New Jersey, USA). Glucose (GPA), triglycerides (TG), and total cholesterol (TC) will be measured by means of a dry analytical methodology in an automated equipment VITROS® 250 (Ortho-Clinical Diagnostics Johnson & Johnson, Rochester, NY, USA).The same equipment will be used to perform liver function tests, albumin, globulins, alkaline phosphatase, lactic dehydrogenase, aspartate aminotransferase, alanine aminotransferase.

Glycosylated hemoglobin. The Glycohemoglobin Pre-Fil of StanbioLab® kit of reagents (Boerne, Texas, USA) will be used. For each standard and sample, the absorbance range will be calculated according to the formula provided by the manufacturer. The conversion factor will be used, and results will be reported as HbA1c. Values between 4.2% and 6.2% will be considered normal.

microRNA determination. For the determination of miRNA, the reagent kits of Quiagen® will be used. The kit miRNeasly Serum/Plasma will be used to obtain the RNA. Once the RNA has been purified from the blood samples, the oligo T retrotranscriptase reaction will be performed using the miScript II RT kit and the buffer miScript HiSpec. Afterwards, the amplification of the miARN of interest will be made in a real time thermocycler with the miScript miRNA polimerase chain reaction (PCR) Array Human Diabetes kit. To visualize amplicons, the investigators will use the miScript SYBR Green PCR kit. Results will be assessed with the software of the real time thermocycler to measure differences in transcription levels. The thermocycler will analyze the increments-decrements in the signals of the selected miARN: miR-320, miR-33a/b, miR-145, miR-335, and miR-124a. The miScript Primer Assay from Quiagen® will be used. As controls of the amplification reactions, the investigators will use mi-rtc as control of the efficiency of the retrotranscriptase and mir-3p from C. elegans as a PCR control.

Statistical analysis. For data processing, version 21.0 of the Statistics Package for the Social Sciences (SPSS, Chicago, Illinois, USA) will be used. For data analysis, descriptive statistics with central tendency will be used, as well as contingency tables. The test for related samples will be used to compare variables in the groups, according to the biochemical markers and gender of participants, Pearson's correlation test will also be used to compare variables among groups and gender. Statistical significance will be set at p ≤ 0.05.

Ethical considerations. The study was submitted for approval to the Research and Ethics Committees of the DACS to be registered at the Research Division of the Universidad Juárez Autónoma de Tabasco, code UJAT-DACS-2015-IA-08. The study complies with the Helsinki Declaration of the World Medical Association. The design complies with the regulations contained in the General Law on Health Research of Mexico.

ELIGIBILITY:
Inclusion Criteria:

* be student in DACS-UJAT
* accept to eat traditional-food

Exclusion Criteria:

* those students being treated for diabetes mellitus
* those students taking lipid-lowering drugs
* those students pregnant
* out of the 20- to 22-year-old range

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Changes on biochemical parameters and selected miRNA | At end 12 week
  The multiple measurements will be aggregate to evaluate the number of participants with abnormal laboratory values pre and post treatment and compare with control.
  Changes in the expression of microRNA selected. The hypothesis are with traditional-type food the biochemical parameters will be lesser than with cafeteria fast-food.
  Adverse events that can occur are hives, nausea and vomiting, abdominal distension, flatulence, diarrhea. It will be compared with the number of adverse events that occur in the control group. Traditional ethnic food is made with local products, especially vegetable. Although these are products that the population has consumed before, they can arise allergy from any product for which will be monitored after each meal.

REFERENCES:
- [Background] Fonseca-Sanchez MA, Perez-Plasencia C, Fernandez-Retana J, Arechaga-Ocampo E, Marchat LA, Rodriguez-Cuevas S, Bautista-Pina V, Arellano-Anaya ZE, Flores-Perez A, Diaz-Chavez J, Lopez-Camarillo C. microRNA-18b is upregulated in breast cancer and modulates genes involved in cell migration. Oncol Rep. 2013 Nov;30(5):2399-410. doi: 10.3892/or.2013.2691. Epub 2013 Aug 22. PMID 23970382
- [Result] Munoz-Cano JM, Cordova-Hernandez JA, del Valle-Leveaga D. [The healthy eating index of new students at an university of Mexico]. Nutr Hosp. 2015 Apr 1;31(4):1582-8. doi: 10.3305/nh.2015.31.4.8401. Spanish. PMID 25795944
- [Result] Munoz Cano JM, Cordova Hernandez J, Mayo H, Boldo Leon X. [Pre-diabetes and diabetes without association with overweight or obesity in Mexican youth]. Arch Latinoam Nutr. 2013 Jun;63(2):148-56. Spanish. PMID 24934071
- [Result] Munoz Cano JM, Aguilar AC, Hernandez JC. Lipid-lowering effect of maize-based traditional Mexican food on a metabolic syndrome model in rats. Lipids Health Dis. 2013 Mar 15;12:35. doi: 10.1186/1476-511X-12-35. PMID 23497051